CLINICAL TRIAL: NCT04826432
Title: Efficacy and Feasibility of Pasireotide to Reduce Clinically Relevant Digestive Leakage After Complete Cytoreductive Surgery (CRS) Plus Hyperthermic Intra-Peritoneal Chemotherapy (HIPEC) for Peritoneal Carcinomatosis - a Phase II Randomized Multicentric Trial
Brief Title: Pasireotide to Reduce Clinically Relevant Digestive Leakage After Complete Cytoreductive Surgery (CRS) Plus Hyperthermic Intra-Peritoneal Chemotherapy (HIPEC) for Peritoneal Carcinomatosis
Acronym: PASIREOCHIP
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: No more experimental drugs available
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-002507-18; 2019/2955 (Other: CSET number)
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Peritoneal Carcinomatosis
MeSH Terms: conditions — Peritoneal Neoplasms | interventions — pasireotide; Saline Waters

STUDY DESIGN:
Intervention Model Description: Randomized Single-blinded, multicentric, placebo controlled phase II comparative trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pasireotide (Experimental): 0.9 mg of pasireotide subcutaneously (s.c.) twice daily (14 doses) every 12 +/- 2 hours
  Interventions: Drug: Pasireotide 0.9 MG/ML
- Placebo (Placebo Comparator): 0.9 ml of saline water s.c. twice daily (14 doses) every 12 +/- 2 hours
  Interventions: Other: Saline water

INTERVENTIONS:
Drug: Pasireotide 0.9 MG/ML — 0.9 mg of pasireotide subcutaneously (s.c.) twice daily (14 doses) every 12 +/- 2 hours
  Arms: Pasireotide
Other: Saline water — 0.9 ml of saline water s.c. twice daily (14 doses) every 12 +/- 2 hours
  Arms: Placebo

SUMMARY:
To assess the efficacy of pasireotide in the reduction of clinically relevant postoperative digestive leakage after CRS plus HIPEC compared to placebo

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged between 18 years and 75 years included
* ECOG (Eastern Cooperative Oncology Group) Performance Status ≤ 2
* Primary (pseudomyxoma peritonei, peritoneal mesothelioma) or Secondary (colorectal or ovarian) peritoneal malignancies
* Curative intent resection obtained by a complete resection according to the Completeness of Cytoreduction score (CC) (CC 0-1) followed by HIPEC Different intraperitoneal drug administration modalities such as neoadjuvant systemic plus simultaneous intraperitoneal and intravenous chemotherapy (NIPS) or pressurized intra-peritoneal aerosol chemotherapy (PIPAC) does not represent exclusion criteria.
* Absence of extra-peritoneal metastatic disease or limited hepatic or lung metastases easily amenable to curative-intent resection or ablation
* Intraoperative Peritoneal Cancer Index (PCI score) ≥ 10
* Visceral resection with at least one digestive anastomosis with or without loop ileostomy or pancreatic or biliary resection.
* Negative serum pregnancy test for women of childbearing potential within 7 days prior to therapy
* Sexually active women of childbearing potential must agree to use a highly effective method of contraception or to abstain from sexual activity during the study and for 3 months after the last study treatment administration. Sexually active males patients must agree to use condom or to abstain from sexual activity during the study and for 3 months after the last study treatment administration. Also, it is recommended their women of childbearing potential partner use a highly effective method of contraception during the same period.
* Patient should understand, sign, and date the written informed consent form prior to any protocol-specific procedures performed. Patient should be able and willing to comply with study visits and procedures as per protocol.
* Patients must be affiliated to a social security system or beneficiary of the same

Exclusion Criteria:

* Macroscopically incomplete surgical resection (CC 2)
* Standard contraindications to pasireotide:

  1. patients with uncontrolled diabetes mellitus or a fasting plasma glucose > 250mg/dl (14 mMol/L)
  2. patients who have congestive heart failure (NYHA Class III or IV), unstable angina, sustained ventricular tachycardia, ventricular fibrillation, clinically significant bradycardia including a corrected QT (QTc) interval longer than 450 msec, advanced heart block or a history of acute myocardial infarction within the six months preceding enrollment
  3. patients with liver disease such as severe hepatic impairment (Child Pugh C), chronic active hepatitis or chronic persistent hepatitis with abnormal coagulation (INR>1.5).
  4. patients with the presence of active or suspected acute or chronic uncontrolled infection
  5. hypersensitivity to somatostatin analogues or any component of pasireotide formulations
  6. patients with uncontrolled hypothyroidism
* Patients participating or who have participated to another study evaluating the effect of a new drug other than pasireotide within 1 month prior to dosing
* Patient who have already participated to this study (a patient can only be included once in the study)
* Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable or will be unable to complete the entire study.
* Women who are pregnant or likely to be so, or who are breastfeeding
* Patient under guardianship or deprived of his liberty by a judicial or administrative decision or incapable of giving its consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2024-02-07 (Actual); Study Completion 2024-02-07 (Actual)

PRIMARY OUTCOMES:
postoperative digestive leakage | 97 days
  The rate of clinically relevant (NCI CTCAE v5 ≥ grade 3) postoperative digestive leakage at 97 days

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, France

IPD SHARING:
Plan to Share IPD: Undecided